CLINICAL TRIAL: NCT01665066
Title: Pharmacokinetic Profile of Toxic Substances and Nicotine in Electronic Cigarettes: a Randomised Cross-over Trial KINECIG
Brief Title: Pharmacokinetic Profile of Toxic Substances and Nicotine in Electronic Cigarettes
Acronym: KINECIG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universita degli Studi di Catania (Other)
Collaborators: Laboratory for Health Protection Research (Unknown)
Responsible Party: Principal Investigator, Riccardo Polosa, Professor of Internal Medicine, Universita degli Studi di Catania
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: KINECIG UNICT 526 /12 (Polosa); Polosa-Caponnetto 2012 (Registry Identifier: Kinecig (Polosa-Caponnetto) 2012)
Record Dates: First submitted 2012-07-23; First posted 2012-08-15 (Estimated); Last update posted 2012-12-13 (Estimated); Status verified 2012-12

CONDITIONS: Tobacco Abuse Smoke
MeSH Terms: interventions — Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Own Brand cigarette (Active Comparator): Smoke Own Brand cigarette, 15 puff of cigarette.
  Interventions: Other: Own Brand cigarette; Other: one high 2,4% nicotine; Other: original 7,4 mg nicotine; Other: nicotine free; Other: Ego 9mg
- One High 2,4% nicotine (Experimental): Smoke electronic cigarette One High 2,4% nicotine for a day, 15 puff of e-cigarette.
  Interventions: Other: Own Brand cigarette; Other: one high 2,4% nicotine; Other: original 7,4 mg nicotine; Other: nicotine free; Other: Ego 9mg
- Original 7,4 mg nicotine (Experimental): Smoke electronic cigarette Original 7,4 mg nicotine for a day. 15 puff of e-cigarette.
  Interventions: Other: Own Brand cigarette; Other: one high 2,4% nicotine; Other: original 7,4 mg nicotine; Other: nicotine free; Other: Ego 9mg
- Nicotine Free (Placebo Comparator): Smoke electronic cigarette nicotine free (15 puff)
  Interventions: Other: Own Brand cigarette; Other: one high 2,4% nicotine; Other: original 7,4 mg nicotine; Other: nicotine free; Other: Ego 9mg
- EGO 9mg (Experimental): Smoke electronic cigarette EGO for a day (15 puff)
  Interventions: Other: Own Brand cigarette; Other: one high 2,4% nicotine; Other: original 7,4 mg nicotine; Other: nicotine free; Other: Ego 9mg

INTERVENTIONS:
Other: Own Brand cigarette — Smoke, 15 puff of, Own Brand cigarettes;
Other: one high 2,4% nicotine — Smoke, 25 puff, of electronic cigarette one high 2,4% nicotine
  Other Names: Categoria electronic cigarette one high 2,4% nicotine
Other: original 7,4 mg nicotine — Smoke, 15 puff, of Categoria electronic cigarette 7,4 mg nicotine
  Other Names: Categoria electronic cigarette 7,4 mg nicotine
Other: nicotine free — smoke, 15 puff, of electronic cigarette nicotine free
  Other Names: categoria electronic cigarette nicotine free "mint".
Other: Ego 9mg — smoke, 15 puff, of electronic cigarette Ego 9 mg
  Other Names: electronic cigarette Ego 9 mg nicotine

SUMMARY:
The aim of the present study is to compare serum nicotine levels of different e-Cigarette strength with usual cigarettes. Serum levels of carcinogenic and toxic substances will be also compared.

DETAILED DESCRIPTION:
The study is randomised cross-over trial designed to compare: 1) serum nicotine levels of four different e-Cigarette strength ; 2) Serum levels of carcinogenic and toxic substances will be also compared. Participants will be requested to abstain from smoking and alcohol from 20:00 on the night before each study day and from food and caffeine for at least 1 h before the session. On arrival at the study centre, carbon monoxide (CO) will be measured in participants' expired breath. If CO will be less than 15 parts per million (ppm), the assigned study treatment will be allocated; however, if CO was > 15 ppm or they will report smoking in the previous 12 h, participants will be rescheduled wherever possible to a subsequent session.

On the first study day, participants will be randomised to use one of five ordered conditions (each separated by 3 day): ENDDs (fourth generation) containing nicotine 2,4%; ENDDs (second generation) containing nicotine 7,4 mg; ENDDs containing nicotine 9 mg; ENDDs nicotine free; their usual cigarette. Additionally participants will be trained to use an electronic cigarette. The following tests will be completed at the each visits: Aldehydes; ROM/TOS; Total thiols; Nicotine; Hydroxypyrene; Cotinine; 1,3-butadiene; Acrylonitrile. After, they will be cannulated and serial venous blood samples for Aldehydes; ROM/TOS; Total thiols; Nicotine will be collected at 0.5, 2, 5, 15, 30 and 60 min after being instructed to take 10 puffs. Additionally, levels of carbon monoxide in exhaled breath (eCO) will be measured 0.5, 2, 5, 15, 30 and 60 min after being instructed to take 10 puffs. At 60 min, after being instructed to take 10 puffs, urine sample for Hydroxypyrene; Cotinine; 1,3-butadiene; Acrylonitrile will be collected. Participants then will leave the study centre with instructions to continue their usual daily activities and to use the study product regularly (for at least 10 hrs) and freely throughout the day. At bedtime and after the puffing chronic phase, when participants will use the study product regularly for at least 10 hrs, urine sample for Hydroxypyrene; Cotinine; 1,3-butadiene; Acrylonitrile will be collected. Participants will be allowed to smoke as they will wish once these measures will be collected and during the 3-day washout period between each study day.

ELIGIBILITY:
Inclusion Criteria:

* 20 regular smokers (smoking ≥ 15 factory-made cigarettes per day for at least the past 10 years and not currently attempting to quit smoking or wishing to do so in the next 30 days, CO > 10 parts per million ) will be recruited from the local Hospital staff in Catania, Italy.

Exclusion Criteria:

* people who reported recent myocardial infarction, angina pectoris or other serious medical conditions (diabetes mellitus, severe allergies, poorly controlled asthma or other airways disease, poorly controlled psychiatric disorders or current chemical dependence other than nicotine) and
* pregnancy,
* breastfeeding,
* blood pressure > 180 mm Hg systolic and/or 100 mm Hg diastolic,
* weight < 45 or > 120 kg, or
* current use of any other smoking cessation medications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-05; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
nicotine pharmacokinetic | 0 sec, 30 second, 2 minutes, 5 minutes, 15 minutes, 30 minutes, 60 minutes
  participants will be cannulated and serial venous blood samples for Nicotine will be collected at 0.5, 2, 5, 15, 30 and 60 min after being instructed to take 10 puffs of cigarette

SECONDARY OUTCOMES:
Serum levels of carcinogenic and toxic substances (Aldehydes; ROM/TOS; Total thiols) | 0 sec, 30 second, 2 minutes, 5 minutes, 15 minutes, 30 minutes, 60 minutes
  Compare serum levels of carcinogenic and toxic substances of "Categoria" electronic cigarettes labelled Original 7,4 mg nicotine , Disposable "Categoria" electronic cigarettes labelled One 2,4% nicotine, Disposable "Categoria" electronic cigarettes labelled nicotine free, electronic cigarettes labelled Ego 9mg nicotine with usual cigarettes.

CONTACTS AND LOCATIONS:
Overall Officials: Riccardo Polosa, MD, Phd, Principal Investigator — University of Catania
Locations (1):
- Centro per la Prevenzione e Cura del Tabagismo, Catania, Catania, Italy

REFERENCES:
- [Result] Goniewicz ML, Kuma T, Gawron M, Knysak J, Kosmider L. Nicotine levels in electronic cigarettes. Nicotine Tob Res. 2013 Jan;15(1):158-66. doi: 10.1093/ntr/nts103. Epub 2012 Apr 22. PMID 22529223